CLINICAL TRIAL: NCT03396796
Title: Modified Vagus Nerve-preserving Versus Conventional Laparoscopic Splenectomy and Azygoportal Disconnection
Brief Title: Modified Vagus Nerve-preserving Laparoscopic Splenectomy and Azygoportal Disconnection
Acronym: ESVLSD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yangzhou University (Other)
Responsible Party: Principal Investigator, Guo-Qing Jiang, Clinical Professor, Yangzhou University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: YZUC-003
Record Dates: First submitted 2018-01-04; First posted 2018-01-11 (Actual); Last update posted 2020-01-22 (Actual); Status verified 2020-01

CONDITIONS: Cirrhosis; Hypertension; Splenectomy; Laparoscopy
Keywords: Vagus nerve; Delayed gastric emptying; Cirrhosis; Hypertension; laparoscopy
MeSH Terms: conditions — Fibrosis; Hypertension; Gastroparesis

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vagus nerve-preserving group (Experimental): Every patient of vagus nerve-preserving group will receive the modified vagus nerve-preserving laparoscopic azygoportal disconnection procedure.
  Interventions: Procedure: Vagus nerve-preserving group
- Conventional group (No Intervention): Every patient of conventional group will receive the conventional laparoscopic azygoportal disconnection procedure.

INTERVENTIONS:
Procedure: Vagus nerve-preserving group — The modified vagus nerve-preserving procedure was performed in the following order: (1) left gastroepiploic vein along greater curvature; (2) the posterior surface of stomach, including the posterior gastric veins; (3) the left lateral surface of the distal esophagus; (4) the left inferior phrenic veins; (5) the posterior surface of the distal esophagus;(6) the anterior surface of the distal esophagus; and (7) the right lateral surface of the distal esophagus. The hepatogastric ligament was conserved. the adherent junction between visceral peritoneum and the right crural diaphragm, and divided it into the lesser omental sac. The left gastric artery and vein and the posterior gastric veins were transected en bloc using a linear laparoscopic vascular stapler.
  Arms: Vagus nerve-preserving group

SUMMARY:
This study aimed to evaluate whether vagus nerve-preserving laparoscopic splenectomy and azygoportal disconnection is effective and safe, and to determine whether a reduction in the incidence of postoperative complications of the digestive system improves postoperative quality of life compared with conventional laparoscopic splenectomy and azygoportal disconnection.

DETAILED DESCRIPTION:
After successful screening the cases of cirrhosis of liver irrespective of the etiology who have non tumor portal vein thrombosis will be enrolled. The baseline parameter will be recorded and the patient will be randomized into either interventional (vagus nerve-preserving laparoscopic splenectomy and azygoportal disconnection) or control (conventional laparoscopic splenectomy and azygoportal disconnection) group. From postoperative day 3, all patients will receive 100 mg oral aspirin enteric-coated tablets (Bayer, Leverkusen, Germany) once daily for 1 year, low-molecular-weight heparin (CS Bio, Hebei, China) subcutaneously (4.100 IU/day) for 5 days, and 25 mg of oral dipyridamole (Henan Furen, Henan, China) thrice daily for 3 months. At months 3, 9, and 12 after operation, electron gastroscopy examination for delayed gastric emptying will be done for all patients. Postoperative complications of the digestive system (including diarrhea, epigastric fullness, bloating, nausea, and vomiting), liver and renal function, and body weight will be recorded at the seventh day, months 1, 3, 6, 9, and 12 after operation. Then one year monitoring will be done in the both groups as per the primary or secondary outcome.

ELIGIBILITY:
Inclusion Criteria:

* A clinical, radiological or histologic diagnosis of cirrhosis of any etiology
* Splenomegaly with secondary hypersplenism
* Bleeding portal hypertension
* No evidence of portal vein system thrombosis by ultrasound evaluation and angio-CT
* Informed consent to participate in the study

Exclusion Criteria:

* Delayed gastric emptying
* Diarrhea
* Hepatocellular carcinoma or any other malignancy,
* Hypercoagulable state other than the liver disease related
* DRUGS- oral contraceptives, anticoagulation or anti-platelet drugs.
* Child - Pugh C
* Recent peptic ulcer disease
* History of Hemorrhagic stroke
* Pregnancy.
* Uncontrolled Hypertension
* Age>75 yrs
* Human immunodeficiency virus (HIV) infection

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-04-09 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Delayed gastric emptying | 1 year
  Proportions of patients who will suffer from delayed gastric emptying in both groups.

SECONDARY OUTCOMES:
Postoperative complications of the digestive system | 1 year
  Proportions of patients who will suffer from postoperative complications of the digestive system in both groups.
Body weight | 1 year
  Proportions of patients who will show improvement in body weight both groups.
Hepatic decompensation | 1 year
  Proportions of patients who will suffer from hepatic decompensation defined as development of ascites, PSE, portal hypertensive bleeding, jaundice, spontaneous bacterial peritonitis, or systemic infection.
Portal vein system thrombosis | 1 year
  Proportions of patients who will suffer from portal vein system thrombosis in both groups.
Hepatocellular carcinoma | 1 year
  Proportions of patients who will suffer from hepatocellular carcinoma in both groups.
Overall survival | 1 year
  Overall survival in both groups.

CONTACTS AND LOCATIONS:
Overall Officials: Dou-Sheng Bai, MD, Study Chair — Clinical Medical College of Yangzhou University; Guo-Qing Jiang, MD, Principal Investigator — Clinical Medical College of Yangzhou University; Ping Chen, MD, Study Director — Clinical Medical College of Yangzhou University
Locations (1):
- Clinical Medical College of Yangzhou University, Yangzhou, Jiangsu, China